CLINICAL TRIAL: NCT01651260
Title: Assessment of the Functionality and Performance of an Endotracheal (ET) Tube Protection Device
Brief Title: Assessment of an Endotracheal Tube Securement Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hollister Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5156-I
Record Dates: First submitted 2012-07-16; First posted 2012-07-27 (Estimated); Results first posted 2015-10-28 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-02

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endotracheal (ET) tube securement device (Other): Single arm study evaluated an experimental ET tube securement device with a bite block.
  Interventions: Other: Experimental ET Tube Securement Device

INTERVENTIONS:
Other: Experimental ET Tube Securement Device — Experimental Hollister device with bite block was substituted for standard-of-care device during the study period.
  Other Names: AnchorFast Guard® ET tube securement device

SUMMARY:
Endotracheal intubation is the translaryngeal placement of a tube into the trachea via the nose or mouth. Endotracheal tubes must be securely fixed to prevent movement, which may result in accidental slippage of the tube into a mainstream bronchus or into the pharynx. Hollister Incorporated is assessing the functionality and performance of an endotracheal tube securement device.

DETAILED DESCRIPTION:
This was a multiple site assessment of the Anchor Fast with enhanced tube protection. Subjects already intubated who required a change of tube-securing device or subjects requiring intubation for greater than 24 hours who meet the inclusion and exclusion criteria were eligible to enroll into the study.The study was open to adult subjects without an existing neck injury who required oral tracheal intubation for greater than 24 hours. Subjects were required to have intact skin on the application site and to be free of facial hair, damaged skin or conditions on the application site (e.g. sunburn, scars, moles or other disfigurations), and significant skin diseases on the application site (e.g. psoriasis, eczema, atopic dermatitis, active cancer) which may have contraindicated participation.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 years of age or older; male or female and requiring oral tracheal intubation.
* Has intact skin on application site.
* Willingly signs or their authorized representative willingly signs the Informed Consent.
* Is qualified to participate in the opinion of the Investigator.

Exclusion Criteria:

* Has an existing neck injury.
* Has protruding upper teeth, without teeth or is unable to wear upper dentures.
* Has facial hair.
* Has clinically significant skin diseases on the application site which may contraindicate participation, including psoriasis, eczema, atopic dermatitis, active cancer.
* Has damaged skin or conditions on the application site which includes sunburn, scars, moles or other disfiguration of the test site.
* Has a known or stated allergy to adhesive bandages, or any of the product types being tested.
* Uses of topical drugs on the application site.
* Uses lotions, creams or oils on the application site.
* Currently is participating in any clinical testing which may affect performance of this device.
* Has been previously intubated with skin irritation or pressure sores surrounding the mouth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Konz, PhD, Study Chair — Hollister Incorporated
Locations (5):
- United States (5):
  - Hartford Hospital, Hartford, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - St. Joseph's Hospitals, Tampa, Florida
  - Legacy Good Samaritan, Portland, Oregon
  - Legacy Salmon Creek Medical Center, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between July 2012 to February 2013 in the ICU setting at 6 hospitals.
Groups:
- Hollister ET Tube Securement Device: Hollister endotracheal tube securement device : Subjects wear one Hollister ET tube securement device until the device either needs to be changed or is no longer required by the subject.
Period: Overall Study
Arm/Group | Hollister ET Tube Securement Device
Started | 65
Completed | 62
Not Completed | 3
Not completed — unable to apply product | 3

BASELINE CHARACTERISTICS:
Population: Complete demographic profiles were obtained for 63 participants
Groups:
- Hollister ET Tube Securement Device: Hollister endotracheal tube securement device: Subjects wear one Hollister ET tube securement device until the device either needs to be changed or is no longer required by the subject.
Arm/Group | Hollister ET Tube Securement Device
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 35
Reason for intubation [Number; unit: participants]
  Respiratory Failure | 55
  Post-operative | 3
  Other | 5

OUTCOME MEASURES:

1. Primary Outcome: Prevention of Damage and/or Occlusion of Endotracheal (ET) Tube During Use
Description: Number of participants with damage of ET tube and Number of participants with occlusion of ET tube
Time Frame: 14 days
Measure: Number; unit: participants
Groups:
- Hollister Endotracheal (ET) Tube Securement Device: Hollister endotracheal tube securement device : Subjects wear one Hollister ET tube securement device until the device either needs to be changed or is no longer required by the subject.
Arm/Group | Hollister Endotracheal (ET) Tube Securement Device
Number analyzed (Participants) | 62
participants
  Damage to ET tube | 0
  Occlusion of ET Tube | 1
Statistical Analysis 1: Comparison: Hollister Endotracheal (ET) Tube Securement Device; Test type: Superiority or Other; Minimum sample size of 60 subjects was required based on the ability of the device to perform at an observed level of non-failure equivalent to an expected upper probability of failure not to exceed 5%; upper probability of failure = .05 — Minimum sample size of 60 subjects was required based on the ability of the device to perform at an observed level of non-failure equivalent to an expected upper probability of failure not to exceed 5%

2. Secondary Outcome: Ease of Use
Description: Likert scale score provided by clinician (1 very difficult, 2 difficult, 3 neither easy nor difficult, 4 easy, 5 very easy);
Time Frame: Between 1 - 14 days
Measure: Number; unit: % rating with score of 4 and 5
Arm/Group | Hollister ET Tube Securement Device
Number analyzed (Participants) | 62
% rating with score of 4 and 5 | 63

ADVERSE EVENTS:
Arm/Group | Hollister ET Tube Securement Device
Serious Adverse Events (participants affected / at risk) | 4/65
Other Adverse Events (participants affected / at risk) | 4/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hollister ET Tube Securement Device (N=65)
Obstruction of ET tube (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Blood oxygen saturation (SpO2) dropped from 100% to 60% due to patient biting ET tube. Unrelated to the device.
Loosened teeth (General disorders) | 1 (1) — Three upper teeth loose. Probably related to device.
Death (General disorders) | 1 (1) — Patient on terminal wean expired with device in place. Unrelated to device.
Death (General disorders) | 1 (1) — Patient on terminal wean expired with device in place. Unrelated to device
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Hollister ET Tube Securement Device (N=65)
Ulcer on tongue (Skin and subcutaneous tissue disorders) | 1/1 (1) — Ulcer on tongue possibly related to device.
Upper lip breakdown (Skin and subcutaneous tissue disorders) | 1/1 (1) — Upper lip ulcer probably related to device.
Wound on upper palette (Skin and subcutaneous tissue disorders) | 1/1 (1) — Wound on upper palette probably related to device.
Bleeding tongue. (Skin and subcutaneous tissue disorders) | 1/1 (1) — Patient forced tongue to opposite side of jaw and bit the tongue. Unrelated to the device.

LIMITATIONS AND CAVEATS:
Adult subjects in respiratory insufficiency in ICU setting were intubated with only four ET tube sizes: 7.0, 7.5, 8.0 and 8.5 mm. No other sizes were represented in the sample population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less